CLINICAL TRIAL: NCT03875404
Title: Transform the Practice: Next-Generation Pre-Operative Targeting for Thalamic DBS in the Treatment of Tremor
Brief Title: Next-Generation Pre-Operative Targeting for Thalamic DBS in the Treatment of Tremor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Erik H. Middlebrooks, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18-010340
Record Dates: First submitted 2019-03-08; First posted 2019-03-14 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Essential Tremor
Keywords: Deep Brain Stimulation
MeSH Terms: conditions — Essential Tremor | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deep Brain Stimulation subjects (Experimental)
  Interventions: Diagnostic Test: Functional MRI

INTERVENTIONS:
Diagnostic Test: Functional MRI — A special type of MRI measuring the metabolic changes that occur within the brain. It may be used to examine the brain's anatomy and determine which parts of the brain are handling critical functions. It helps identify important language and movement control areas in the brain.

SUMMARY:
Researchers are investigating improved methods of targeting deep brain stimulators for treatment of essential tremor relying on brain connectivity measures derived from MRI.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of refractory essential tremor scheduled for unilateral thalamic deep brain stimulator placement
* Age ≥ 18 years

Exclusion Criteria:

* Prior deep brain stimulator, stereotactic radiosurgery, or focused ultrasound procedure for treatment of tremor
* Presence of concomitant movement disorder (e.g. Parkinson's disease, dystonia, etc.)
* Known pre-existing structural brain abnormality (e.g, infarction, tumor, prior brain surgery, etc.)
* Contraindication to 3 Tesla brain MRI (e.g. incompatible implanted device)
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-02-12 (Actual)

PRIMARY OUTCOMES:
Change in tremor rating score | One year
  Fahn, Tolosa, Marin Tremor Rating Scale 1-9 Tremor (rate tremor)
  0 = None
  1. = Slight.
  2. = Moderate amplitude.
  3. = Marked amplitude
  4. = Severe amplitude
  0 = Normal
  1. = Mildly abnormal.
  2. = Moderately abnormal.
  3. = Marked abnormal.
  4. = Severely abnormal.

CONTACTS AND LOCATIONS:
Overall Officials: Erik H Middlebrooks, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials